CLINICAL TRIAL: NCT06537115
Title: Clinical Intervention of Idecalcitol Combined With Whey Protein Powder and Exercise for Sarcopenia：a RCT Trial
Brief Title: Clinical Intervention of Idecalcitol Combined With Whey Protein Powder and Exercise for Sarcopenia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2024041
Record Dates: First submitted 2024-07-28; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; intervention; idecalcitol; whey protein powder; exercise
MeSH Terms: conditions — Sarcopenia; Motor Activity | interventions — Exercise; eldecalcitol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Other): After enrollment, professional doctors will conduct a comprehensive assessment of their basic conditions and provide routine interventions, mainly including basic nutrition intervention program guidance, progressive resistance exercise intervention program guidance, safety protection advice, and symptomatic treatment for different complications, with a total intervention period of 24 weeks.
  Interventions: Behavioral: exercise
- experimental group 1 (Other): On the basis of the control group, whey protein powder was given to supplement for 12 weeks.60 grams of protein per day is taken in three divided doses for 12 consecutive weeks. Attention should be paid to monitoring liver and kidney function, and the dosage of protein powder should be adjusted according to the condition of the patient.
  Interventions: Behavioral: exercise; Dietary Supplement: whey protein powder
- experimental group 2 (Other): On the basis of the control group, whey protein powder and eldecalcitol were given for supplementation for 12 weeks.
  (Supplementing whey protein powder: The protein intake is 60 grams per day, taken in three divided doses for 12 consecutive weeks. Attention should be paid to monitoring liver and kidney function, and the dosage of protein powder should be adjusted according to the condition of the patient.
  Supplementing eldecalcitol: eldecalcitol soft gel capsules are taken at an oral dose of 0.75μg once a day for 12 consecutive weeks.)
  Interventions: Behavioral: exercise; Dietary Supplement: whey protein powder; Drug: Eldecalcitol

INTERVENTIONS:
Behavioral: exercise — progressive resistance exercise
Dietary Supplement: whey protein powder — The protein intake is 60 grams per day, taken in three divided doses for 12 consecutive weeks. Attention should be paid to monitoring liver and kidney function, and the dosage of protein powder should be adjusted according to the condition of the patient.
  Arms: experimental group 1; experimental group 2
Drug: Eldecalcitol — Eldecalcitol soft gel capsules are taken at an oral dose of 0.75μg once a day for 12 consecutive weeks.
  Arms: experimental group 2

SUMMARY:
This clinical trial is a multicenter, single-blind, prospective, randomized controlled clinical application study. Subjects who met the trial criteria and signed the informed consent form were randomly divided into a control group, an experimental group 1, and an experimental group 2. After enrollment, the control group underwent a comprehensive assessment of their underlying conditions by professional physicians and received routine interventions, including basic nutritional intervention program guidance, progressive resistance exercise intervention program guidance, safety precautions, and symptomatic treatment for different complications, for a total intervention period of 24 weeks. The experimental group 1, in addition to the interventions provided to the control group, received whey protein powder supplementation for 12 weeks. The experimental group 2, on the other hand, received both whey protein powder and eldecalcitol supplementation on top of the interventions given to the control group, also for 12 weeks. The entire intervention period lasted for 24 weeks. Through regular general assessments, blood tests, measurements of muscle mass, muscle strength, and physical function, as well as analyses of negative adverse events, statistical methods were employed to evaluate the safety and efficacy of the comprehensive intervention methods for sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 or above;

  * Meeting the diagnostic criteria for sarcopenia according to the definition of AWGS; ③ Able to walk, willing to accept a comprehensive intervention plan, and guarantee to complete the treatment course; ④ Both patients and their families agree to participate in this study and sign the informed consent form.

Exclusion Criteria:

* Resting systolic blood pressure > 200 mmHg or resting diastolic blood pressure > 100 mmHg;

  * Severe heart disease: moderate to severe aortic valve stenosis, acute pericarditis, acute myocarditis, myocardial infarction, uncontrollable arrhythmia;

    * Acute stroke within the past 2 years;

      * Severe airway obstruction;

        * Lower limb fractures in the past 1 year or upper limb fractures in the past 6 months;

          * Hypercalcemia (corrected albumin serum calcium > 2.60 mmol/L);

            * Active malignant tumors; ⑧ Chronic kidney disease stages 5;

              * Mental illness or severe cognitive impairment;

                * Long-term immobilization; ⑪ Other diseases that may interfere with the evaluation of muscle mass, muscle strength, and physical function; ⑫ Unable to cooperate with treatment due to other reasons; ⑬ Life expectancy less than 6 months.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-06-16 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
muscle mass | up to 24 weeks
  The DXA equipment is used to detect the muscle mass.

SECONDARY OUTCOMES:
Grip strength | up to 24 weeks
  Using a spring dynamometer, stand upright with the elbow joint fully extended, and use the muscle strength of the dominant hand to record the maximum reading (in kg) from three trials.
6-meter walking speed | up to 24 weeks
  Record the time required to walk 6 meters from the starting point at a normal speed without decelerating, and use the average result of 3 trials as the recorded walking speed (in m/s).
incidence of adverse reactions | up to 24 weeks
  The number of patients with adverse events within a unit time / the total number of patients in the experimental or control group during the same period * 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Jianfang Ni, bachelor, Principal Investigator — Zhejiang Provincial People's Hospital
Locations (5):
- China (5):
  - The First People's Hospital of Chun'an County, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Huzhou Nanxun District People's Hospital, Huzhou, Zhejiang
  - Xianju People's Hospital, Taizhou, Zhejiang
  - Dinghai Central Hospital of Zhoushan City, Zhoushan, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
The raw data will be uploaded to the ResMan platform for raw data sharing, whose website is: http://www.medresman.org.cn/.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the completion of the study,for 3 years
Access Criteria: username and password
URL: http://www.medresman.org.cn/.

REFERENCES:
- [Background] Chen LK, Woo J, Assantachai P, Auyeung TW, Chou MY, Iijima K, Jang HC, Kang L, Kim M, Kim S, Kojima T, Kuzuya M, Lee JSW, Lee SY, Lee WJ, Lee Y, Liang CK, Lim JY, Lim WS, Peng LN, Sugimoto K, Tanaka T, Won CW, Yamada M, Zhang T, Akishita M, Arai H. Asian Working Group for Sarcopenia: 2019 Consensus Update on Sarcopenia Diagnosis and Treatment. J Am Med Dir Assoc. 2020 Mar;21(3):300-307.e2. doi: 10.1016/j.jamda.2019.12.012. Epub 2020 Feb 4. PMID 32033882
- [Background] Cruz-Jentoft AJ, Sayer AA. Sarcopenia. Lancet. 2019 Jun 29;393(10191):2636-2646. doi: 10.1016/S0140-6736(19)31138-9. Epub 2019 Jun 3. PMID 31171417
- [Background] Maeda K, Imatani J, Moritani S, Kondo H. Effects of eldecalcitol alone or a bone resorption inhibitor with eldecalcitol on bone mineral density, muscle mass, and exercise capacity for postmenopausal women with distal radius fractures. J Orthop Sci. 2022 Jan;27(1):139-145. doi: 10.1016/j.jos.2020.11.009. Epub 2020 Dec 19. PMID 33349543